CLINICAL TRIAL: NCT05876234
Title: The Predictive Value of the Progesterone Level on the Day of Embryo Transfer in Cryo Cycles
Brief Title: The Predictive Value of Progesterone
Acronym: PFRET
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0223
Record Dates: First submitted 2023-05-08; First posted 2023-05-25 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Subfertility
Keywords: progesterone; embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate a 5 ng/ml serum progesterone (P4) threshold policy for the addition of subcutaneous (SC) P4 in artificially prepared frozen embryo transfer cycles treated with vaginal P4. We assess whether the addition of SC P4 rescues cycles with serum P4 <5 ng/ml and we study the impact of not supplementing cycles with serum P4 >5 ng/ml by comparing them with serum P4 cycles above the conventionally proposed cut-off of 10 ng/ml.

ELIGIBILITY:
* Embryo transfer between March 1st 2021 and March 31st 2023
* Determination of progesterone on the day of embryo transfer

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Treated at Ghent University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 11 to 13 weeks after last menstruation
  Fetal heart beat at ultrasound

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6 to 8 weeks after last menstruation
  Ultrasound visualisation of the gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Stoop, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital - Department of Reproductive Medicine, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided